CLINICAL TRIAL: NCT06768164
Title: Health-Related Quality Of Life After Partial Gastrectomy for Gastric Cancer: Comparison of Reconstruction by Billroth II or Roux-en-Y. A Randomized, Comparative, Multicentric, Single-blinded Study
Brief Title: Quality of Life After Billroth II or Roux-en-Y for Gastric Cancer
Acronym: BYQoL-GC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP210355; 2022-A00730-43 (Other: ID-RCB)
Record Dates: First submitted 2024-09-24; First posted 2025-01-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Gastric (Cardia, Body) Cancer
Keywords: gastric cancer; gastrectomy
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms | interventions — Anastomosis, Roux-en-Y

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Billroth 2 (B2) (Experimental)
  Interventions: Procedure: Billroth 2 (B2)
- Roux-En-Y (REY) (Experimental)
  Interventions: Procedure: Roux-En-Y (REY)

INTERVENTIONS:
Procedure: Billroth 2 (B2) — B2 technique requires a single anastomosis (gastro-jejunostomy) after distal gastrectomy
  Arms: Billroth 2 (B2)
Procedure: Roux-En-Y (REY) — REY technique requires 2 anastomoses (gastro-jejunostomy and entero-enterostomy) after distal gastrectomy
  Arms: Roux-En-Y (REY)

SUMMARY:
The treatment of a local distal gastric cancer remains surgical before or after chemotherapy. Partial gastrectomy is recommended for distal location cancer The recommendations for restoring continuity are less evident. There are two main techniques: the Roux-En-Y (REY) requiring 2 anastomoses (gastro-jejunostomy and entero-enterostomy) and the Billroth 2 (B2) with a single anastomosis (gastro-jejunostomy). The choice remains matter of debate.

There was no difference on the global health status score from the QLQ-C30 questionnaire. However, the health-related quality of life (HRQoL) was significantly improved only in the REY group between pre- and post-gastrectomy. A significant difference for endoscopic gastritis in favor of the REY group was reported.

The purpose of this study is to determine which surgical technique improve the health related quality of life after distal gastrectomy.

DETAILED DESCRIPTION:
The realization of REY suggests an improvement of the HRQoL after distal gastric resection in comparison to the B2 anastomosis justifying the need of a RCT on the topic. Moreover, the REY could improve the gastro-intestinal symptoms and gastritis. The investigators hypothesize that the REY intervention after distal gastrectomy will improve HRQoL for 3 targeted dimensions of the EORTC QLQ-OG25 questionnaire (eating, reflux, pain and discomfort) in patients with gastric cancer.

All patients with a distal gastric cancer treated in curative intent by surgery with distal gastrectomy should be included. The choice of this population belongs in the fact that no reconstruction according billroth2 are performed for other gastric cancer requiring a total gastrectomy. Therefore, all patients treated by total gastrectomy need to be excluded. Secondly, the increase in survival of this population in the past decade araising to 75% at 5 years allows investigators to question the quality of life after surgery.

The anastomosis is realized with the proximal jejunum without entero-enterostomy in the first 70 cm after the angle of Treitz. The gastrojejunostomy could be ante-colic or trans-mesocolic. The anastomosis could be performed according the surgeon decision (mechanical or handsewn, isoperistaltic or anisoperistaltic).

The length of jejunum of the Y section needs to be at least 60 cm. The Roux-en-Y anastomosis could be antecolic or transmesocolic. The anastomosis could be realized according the surgeon decision (mechanical or handsewn, isoperistaltic or anisoperistaltic).

The choice between these two techniques will not add an increased risk to the patient since they are both recommended by national guidelines, they are both performed as standard care and there is no difference in Quality of Life at long term.

During surgery:

* A complete exploration of abdominal cavity is realized to avoid presence of peritoneal metastasis. This exploration is allowed by laparoscopy or open surgery
* The gastric tumor permits to realize R0 resection with 5 cm of resection margin according to the subtotal gastric resection on the line between the right side of gastro-esophageal junction and the end of the left gastro-omental artery
* In case of Linitis plastica, realization of anatomopathological examination of proximal margin without sign of tumoral involvement to access to randomization The type of surgery (B2 or REY) will be then determined by randomization

Interventions added for the research are:

* Randomization : the randomization will be realized by the investigator team
* One endoscopy at 1 year of follow-up after surgery
* Quality of Life questionnaires (EORTC QLQ-C30 and QLQ-OG25) at baseline, 3 months, 6 months, 1 year and 2 years of follow-up after surgery

Expected benefits for the participants: Improve HRQoL after distal gastrectomy. Patients will not be exposed to a specific risk as the two methods of reconstruction are described and used in the routine.

The design of the study (without excessive invasive exam) and the routine care monitoring associated to a better HRQoL evaluation compared to the "classic" post-operative follow-up of patient will help patient decision to participate to the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years, men or women
* Patients treated for adenocarcinoma of the antrum accessible to a surgical treatment with curative intent by distal gastrectomy. If patients present a linitis plastica, negative proximal and distal margin will be evaluated at the beginning of the surgery before randomization in order to perform a R0 resection
* Patients with a registration in a national health care system (CMU included) (registered or being a beneficiary of such a scheme)
* Patients able to understand and fulfill questionnaires in French language
* Patients having given their written informed consent prior to participation in the study

Exclusion Criteria:

* Patients with preoperative peritoneal metastasis or distant metastasis
* Palliative surgery patients
* Patients under tutorship or curatorship and protected adults
* Patients on AME (Aide Médicale de l'Etat = State Medical Assistance)
* Patients deprived of liberty by judicial or administrative decision and patients under psychiatric care (admitted to a health or social care establishment)
* Patients unable to give their consent
* Pregnant or breastfeeding women
* Women of childbearing age without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
HRQol with 3 targeted dimensions | One year post-surgery
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, OesophagoGastric 25 (EORTC QLQ-OG25) at 1 year post surgery with 3 targeted dimensions : eating, reflux, pain and discomfort. Health-related Quality of life (HRQoL) will be considered as being improved in one arm if at least one of the 3 targeted dimensions is significantly improved without a significantly deterioration for the other 2 targeted dimensions :
  * Eating restrictions : [0-100].
  * Reﬂux : [0-100].
  * Pain and discomfort : [0-100]. If high scores = more problems.

SECONDARY OUTCOMES:
Other EORTC QLQ-OG25 dimensions | Baseline, 3 months, 6 months, 1 year and 2 years post-surgery
  Other dimensions of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, OesophagoGastric 25 (EORTC QLQ-OG25) questionnaire :
  * Dysphagia : [0-100].
  * Odynophagia : [0-100].
  * Anxiety : [0-100]. If high scores = more problems.
Other HRQoL dimensions | Baseline, 3 months, 6 months, 1 year and 2 years post-surgery
  Other dimensions of the HRQoL measured with the EORTC QLQ-C30 ( European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaires, Core 30) questionnaire will be described at baseline, 3 months, 6 months, 1 year and 2 years post-surgery :
  * Physical function : [0-100].
  * Role function : [0-100].
  * Emotional function : [0-100].
  * Cognitive function : [0-100].
  * Social function : [0-100].
  * Overall quality of life : [0-100]. For these dimensions above if high score = better function.
  * Pain : [0-100].
  * Fatigue : [0-100].
  * Nausea and vomiting : [0-100]. For these dimensions above if high score = more problems.
Longitudinal changes of each HRQoL dimension | The long-term HRQoL (EORTC QLQ-OG25 questionnaire) after surgery for gastric cancer at 2 years
  - The long-term HRQoL after surgery for gastric cancer at 2 years
Longitudinal changes of each HRQoL dimension | et The long-term HRQoL (EORTC QLQ-C30 questionnaire) after surgery for gastric cancer at 2 years
  The long-Term HRQoL after surgery for gastric cancer at 2 years
The long-term HRQoL after surgery for gastric cancer at 2 years | 2 years post-surgery
  The long-term HRQoL after surgery for gastric cancer at 2 years (EORTC QLQ-C30 )
The long-term HRQoL after surgery for gastric cancer at 2 years | 2 years post-surgery
  The long-term HRQoL after surgery for gastric cancer at 2 years (EORTC QLQ-OG25)
The post-operative morbidity rates at 90 days | 90 days post-surgery
  The postoperative morbidity at 90 days will be measured with the several following complications: Surgical site infection / leakage, gastroparesis, gastro-intestinal occlusion, stasis syndrome, dumping syndrome, ulcerative pathology
The post-operative morbidity rates at 1 year | 1 year post-surgery
  The postoperative morbidity at 1 year post surgery will be measured with the several following complications: Surgical site infection / leakage, gastroparesis, gastro-intestinal occlusion, stasis syndrome, dumping syndrome, ulcerative pathology
The endoscopic biliary reflux rate and gastritis at 1 year post surgery | 1 year post-surgery
  The biliary reflux and gastritis will be assessed by endoscopy at 1 year post-surgery
The rate of proton pump inhibitor (PPI) use at 3 months, 6 months, 1 year and 2 years post-surgery | 3 months, 6 months, 1 year and 2 years post-surgery
  The use of PPI will be measured by taking PPI in the past week at 3 months, 6 months, 1 year and 2 years post-surgery
The survival at 1 year | 1 year post-surgery
  The survival at 1 year post-surgery will be recorded by OS and DFS rate. DFS, defined as the time from surgery and locoregional recurrence, occurrence of distant metastases or second gastric cancer, or death (all causes) or the date of the last follow-up, at which point data will be censored.
  OS, defined as the time from surgery to the death from any cause or the date of the last follow-up, at which point data will be censored.
The survival at 2 years | 2 years post-surgery
  The survival at 2 years post-surgery will be recorded by OS and DFS rate. DFS, defined as the time from surgery and locoregional recurrence, occurrence of distant metastases or second gastric cancer, or death (all causes) or the date of the last follow-up, at which point data will be censored.
  OS, defined as the time from surgery to the death from any cause or the date of the last follow-up, at which point data will be censored.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre CHALLINE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint-Antoine, Paris, France